CLINICAL TRIAL: NCT04261842
Title: Identifying the Core Content of Military Identity for Psychological Understanding
Brief Title: Military Identity Project
Status: Completed | Type: Observational
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); University of Rochester (Other); San Antonio Military Medical Center (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency); Womack Army Medical Center (U.S. Federal Agency); Tripler Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FDG20180009E; HU00011820041 N18-B07 (Other Grant/Funding Number: Uniformed Services University of the Health Sciences)
Record Dates: First submitted 2020-01-31; First posted 2020-02-10 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Military Identity; Self-schemas; Psychological Well-being
Keywords: Military Identity; Military psychological health; Active Duty; Well-being; Readiness; Self and Identity; Self-Schemas
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Military Identity Project is an exploration of military identity in Active Duty Service Members of the Army, Navy, Air Force & Marine Corps. The purpose of this project is to discover common identity attributes shared by active duty members across Service branches and to see if specific traits are related to levels of well-being and resilience.

DETAILED DESCRIPTION:
Rationale: Psychological health (PH) disorders continue to be the highest consumer of inpatient bed days and are in the top 10 diagnoses for Active Duty Service Members (ADSM) lost duty days and appointment utilization. Cognitive therapies (CT) are the evidence-based choice for PH conditions. Little is known about the cognitive contents of Military Identity (MI) and the potential for identifying specific cognitive vulnerabilities and resources common in ADSMs. Understanding the role of MI in common military PH conditions can inform the development of new military-specific clinical strategies for CTs.

Study Objective: To validate findings from a pilot Military Identity (MI) study utilizing a self-schema model to determine core cognitive contents of MI and to explore relationships between MI and psychological well-being (PWB).

Specific Aims:

Aim 1: Describe the core cognitive content of MI in active duty service members.

Aim 2: Examine the effect of MI on information processing response times.

Aim 3: Explore the relationship between MI and self-perceived psychological well-being scores.

Design: A descriptive cross-sectional mixed methods content analysis and a four-group information processing paradigm will be utilized to investigate a stratified sample of ADSMs across Joint Services (25% sample from each Army, Navy, Air Force, Marine).

Methods: Open-Ended and Closed-Ended Identity Attribute Tasks will be used to explore MI content as well as a 60 attribute response time task along with a demographic questionnaire, Inclusion of In-group in Self Scale, and Ryff's PWB Scales. All measures will be collected via computerized software program developed by Harvard's Project Implicit.

Dissemination of Results: Results from the study will be disseminated through publications, poster and/or podium presentations at professional annual conferences such as the American Psychological Association (APA), Military Health Systems Research Symposium, Association of Military Surgeons United States (AMSUS), and Tri-Service Nursing Research Program (TSNRP). Manuscripts will be submitted for publication to appropriate journals such as Military Psychology, Military Behavioral Health, and Military Medicine.

ELIGIBILITY:
Inclusion Criteria:

* An active duty member of the US Army, US Air Force, US Marine Corps, US Navy
* Willing to complete the online identity tasks requiring approximately 45 minutes

Exclusion Criteria:

* Civilian
* Guard or Reserve Service Members
* U.S. Public Health Service Member
* U.S. Coast Guard Service Member

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population of interest includes a stratified self-selected sample of ADSM participants (25% USA, 25% USAF, 25% USMC, 25% USN). Recruitment will be primarily through online forums with facilitation championed from five recruitment hubs at: 1) David Grant Medical Center (USAF) serving over 10K ADSM, 2) 59th Medical Wing, (USAF) serving over 60K ADSM, 3) Walter Reed National Military Medical Center, (USN) serving over 3.5K ADSM, 4) Womack Army Medical Center (USA) serving 50K ADSM. and 5) Marine Corps Base Hawaii (USMC), home to the majority of the 5,300 Marines stationed on Oahu. The study is site agnostic as it will be conducted in a virtual environment hosted by Harvard's Project Implicit virtual laboratory, therefore any ADSM who meets the inclusion criteria is eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Open-ended Identity Attribute Task (Task 1) | 15 minutes
  Participants will enter up to 9 attributes that represent how they think about themselves as a military member and using an 11-point scale rate each attribute according to: Self-descriptiveness (How much does this attribute really describe me?), Importance (How important is this attribute to who I am as a military member?) and, Valence (How positive or negative do I consider this attribute in myself?).
Identity Attribute Response Time Task (Task 2) | 3 minutes
  The Response Time task will involve participants striking specific keys on the keyboard to endorse or reject 70 pre-determined attributes (10 practice attributes; 60 randomized experimental attributes) as self-descriptive.
Demographic Questions (Task 3) | 2 minutes
  The participant will respond to six demographic items: gender, Service branch, rank, active duty service time, number of deployments, and whether raised in a military family.
Inclusion of In-group in the Self Scale (Task 4) | 1-2 minutes
  The Inclusion of In-group in the Self Scale (IIS) is a single-item measure that is adapted easily and administered quickly for studies involving membership in many different groups. The scale of 1 to 7 is represented by seven pairs of circles representing level of identification with the military; participants will be asked to choose the pair of circles that best represents their own level of identification with the military. The pair of circles labeled "1" (no overlap) represents the lowest level of identification with the military. The pair labeled "7" (almost complete overlap) represents the highest level of identification with the military. The score represents a self-report of a participant's level of identification with a group, and is not by itself indicative of a better or worse outcome.
Closed-ended Identity Attribute Task (Task 5) | 10 minutes
  The Closed-ended Identity Attribute Task (CIAT) provides a list of 60 attributes generated through methods established in the social psychological sciences. Using an 11-point scale, the participant must rate each attribute according to: Self-descriptiveness (How much does this attribute really describe me?), Importance (How important is this attribute to who I am as a military member?) and, Valence (How positive or negative do I consider this attribute in myself?). The CIAT uses the same 60 attributes presented as experimental stimuli in the Identity Attribute Response Time Task (Task 2).
Ryff Scales of Psychological Well-being (Task 6) | 10 minutes
  The Ryff Scales of Psychological Well-being (PWB) is comprised of six 9-item scales (54 total items) of psychological well-being constructed to measure the dimensions of autonomy, environmental mastery, personal growth, positive relations, purpose in life and self-acceptance. Participants will respond to statements using a scale of 1 (Strongly Disagree) to 6 (Strongly Agree). Scores from the 54 items are summed; the higher the total score = the higher the PWB.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie A Migliore, PhD, Principal Investigator — David Grant USAF Medical Center
Locations (1):
- David Grant USAF Medical Center, Travis Air Force Base, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Association of Nurse Practitioners. (2015). NP Facts. Www.Aanp.Org, 78711. Retrieved from https://www.aanp.org/images/documents/about-nps/npfacts.pdf
- [Background] Andersen, B. L., & Cyranowski, J. M. (1994). Women's sexual self-schema. Journal of Personality and Social Psychology. http://doi.org/10.1037/0022-3514.67.6.1079
- [Background] Anderson NH. Likableness ratings of 555 personality-trait words. J Pers Soc Psychol. 1968 Jul;9(3):272-9. doi: 10.1037/h0025907. No abstract available. PMID 5666976
- [Background] Armed Forces Health Surveillance Branch. Absolute and relative morbidity burdens attributable to various illnesses and injuries, active component, U.S. Armed Forces, 2016. MSMR. 2017 Apr;24(4):2-8. No abstract available. PMID 28488875
- [Background] Baayen, H. R., & Milin, P. (2010). Analyzing reaction times. International Journal of Psychological Research, 3(2).
- [Background] Beck AT. The evolution of the cognitive model of depression and its neurobiological correlates. Am J Psychiatry. 2008 Aug;165(8):969-77. doi: 10.1176/appi.ajp.2008.08050721. Epub 2008 Jul 15. PMID 18628348
- [Background] Berghaus, P. T., & Cartagena, N. L. (2013). Developing good soldiers: The problem of fragmentation within the Army. Journal of Military Ethics, 12(4), 287-303. http://doi.org/10.1080/15027570.2013.869389
- [Background] Brewin CR, Garnett R, Andrews B. Trauma, identity and mental health in UK military veterans. Psychol Med. 2011 Aug;41(8):1733-40. doi: 10.1017/S003329171000231X. Epub 2010 Dec 14. PMID 21144125
- [Background] Brewin CR. Understanding cognitive behaviour therapy: A retrieval competition account. Behav Res Ther. 2006 Jun;44(6):765-84. doi: 10.1016/j.brat.2006.02.005. Epub 2006 Apr 18. PMID 16620779
- [Background] Corte C, Stein KF. Self-cognitions in antisocial alcohol dependence and recovery. West J Nurs Res. 2007 Feb;29(1):80-99. doi: 10.1177/0193945906295480. PMID 17228062
- [Background] Cyranowski JM, Aarestad SL, Andersen BL. The role of sexual self-schema in a diathesis-stress model of sexual dysfunction. Appl Prev Psychol. 1999;8(3):217-228. doi: 10.1016/S0962-1849(05)80078-2. PMID 19587834
- [Background] Daley, J. G. (1999). Understanding the military as an ethnic identity. Social work practice in the military, 291-303.
- [Background] Dalgleish T. Cognitive approaches to posttraumatic stress disorder: the evolution of multirepresentational theorizing. Psychol Bull. 2004 Mar;130(2):228-60. doi: 10.1037/0033-2909.130.2.228. PMID 14979771
- [Background] Danish SJ, Antonides BJ. The challenges of reintegration for service members and their families. Am J Orthopsychiatry. 2013 Oct;83(4):550-8. doi: 10.1111/ajop.12054. PMID 24164527
- [Background] Demers, A. (2011). When Veterans return: The role of community in reintegration. Journal of Loss and Trauma, 16(2), 160-179. http://doi.org/10.1080/15325024.2010.519281
- [Background] Deployment Health Clinical Center. (2017). Mental health disorder prevalence among active duty service members in the Military Health System, Fiscal Years 2005 - 2016 prepared by the Deployment Health Clinical Center, (January).
- [Background] Disner SG, Beevers CG, Haigh EA, Beck AT. Neural mechanisms of the cognitive model of depression. Nat Rev Neurosci. 2011 Jul 6;12(8):467-77. doi: 10.1038/nrn3027. PMID 21731066
- [Background] Dobson KS. The science of CBT: toward a metacognitive model of change? Behav Ther. 2013 Jun;44(2):224-7. doi: 10.1016/j.beth.2009.08.003. Epub 2011 Jun 6. PMID 23611072
- [Background] Dozois, D., & Dobson, K. (2003). The structure of the self-schema in clinical depression: Differences related to episode recurrence. Cognition & Emotion, 17(6), 933-941. http://doi.org/10.1080/02699930244000363
- [Background] Dozois DJ, Bieling PJ, Patelis-Siotis I, Hoar L, Chudzik S, McCabe K, Westra HA. Changes in self-schema structure in cognitive therapy for major depressive disorder: a randomized clinical trial. J Consult Clin Psychol. 2009 Dec;77(6):1078-88. doi: 10.1037/a0016886. PMID 19968384
- [Background] Dozois DJ, Dobson KS. Information processing and cognitive organization in unipolar depression: specificity and comorbidity issues. J Abnorm Psychol. 2001 May;110(2):236-46. doi: 10.1037//0021-843x.110.2.236. PMID 11358018
- [Background] Evans, D., Dalgleish, T., Dudas, R. B., Denman, C., Howard, M., & Dunn, B. D. (2015). Examining the shared and unique features of self-concept content and structure in borderline personality disorder and depression. Cognitive Therapy and Research, 39(5), 613-626. http://doi.org/10.1007/s10608-015-9695-3
- [Background] Foa EB, Gillihan SJ, Bryant RA. Challenges and Successes in Dissemination of Evidence-Based Treatments for Posttraumatic Stress: Lessons Learned From Prolonged Exposure Therapy for PTSD. Psychol Sci Public Interest. 2013 May;14(2):65-111. doi: 10.1177/1529100612468841. PMID 25722657
- [Background] Franke, V. (1999). Preparing for Peace. Miltary Identity, Value Orientations, and Professional Military Education. Igarss 2014. http://doi.org/10.1007/s13398-014-0173-7.2
- [Background] Ghosh VE, Gilboa A. What is a memory schema? A historical perspective on current neuroscience literature. Neuropsychologia. 2014 Jan;53:104-14. doi: 10.1016/j.neuropsychologia.2013.11.010. Epub 2013 Nov 23. PMID 24280650
- [Background] Gilboa A, Moscovitch M. Ventromedial prefrontal cortex generates pre-stimulus theta coherence desynchronization: A schema instantiation hypothesis. Cortex. 2017 Feb;87:16-30. doi: 10.1016/j.cortex.2016.10.008. Epub 2016 Oct 31. PMID 27890323
- [Background] Government Accountability Office. (2016). Defense health care: DOD is meeting most mental health care access standards , but it needs a standard for follow- up appointments.
- [Background] Green G, Emslie C, O'Neill D, Hunt K, Walker S. Exploring the ambiguities of masculinity in accounts of emotional distress in the military among young ex-servicemen. Soc Sci Med. 2010 Oct;71(8):1480-8. doi: 10.1016/j.socscimed.2010.07.015. Epub 2010 Aug 5. PMID 20739109
- [Background] Griffith, J. (2011). Reserve identities: What are they? And do they matter? An empirical examination. Armed Forces & Society, 37(4), 619-635. http://doi.org/10.1177/0095327X10382213
- [Background] Griffith, J., & Vaitkus, M. (2013). Perspectives on suicide in the Army National Guard. Armed Forces & Society, 39(4), 628-653. http://doi.org/10.1177/0095327X12471333
- [Background] Gillihan, S. J., Conklin, P., & Foa, E. B. (2014). Dissemination and implementation of evidence-based treatments. The Wiley handbook of anxiety disorders, 1228-1241.
- [Background] Harris, K., Gringart, E., & Drake, D. (2013). Military retirement: Reflections from former members of Special Operations Forces. Identity, 10(3), 97-112. Retrieved from http://www.army.gov.au/Our-future/LWSC/Our-publications/Australian-Army-Journal/~/media/Files/Our future/LWSC Publications/AAJ/2013Winter/AustralianArmyJournal_V10N3Winter_Identity-MilitaryRetirement.pdf
- [Background] Jobson L, O'Kearney R. Cultural differences in personal identity in post-traumatic stress disorder. Br J Clin Psychol. 2008 Mar;47(Pt 1):95-109. doi: 10.1348/014466507X235953. PMID 17708833
- [Background] Johansen, R. B., Laberg, J. C., & Martinussen, M. (2013). Military identity as predictor of perceived military competence and skills. Armed Forces & Society, (May). http://doi.org/10.1177/0095327X13478405
- [Background] Kelley PW, Kenny D, Donley R. Experiences of vulnerability and uncertainty during the Iraq and Afghanistan wars: Stories of wounded service members and the nurses who cared for them. Nurs Outlook. 2017 Sep-Oct;65(5S):S71-S80. doi: 10.1016/j.outlook.2017.08.007. Epub 2017 Aug 12. PMID 28886867
- [Background] Kendzierski, D. (1988). Self-schemata and exercise. Basic and Applied Social Psychology, 9(1), 45-59. http://doi.org/10.1207/s15324834basp0901_4
- [Background] Kendzierski D. Exercise self-schemata: cognitive and behavioral correlates. Health Psychol. 1990;9(1):69-82. doi: 10.1037//0278-6133.9.1.69. PMID 2323330
- [Background] Kihlstrom, J. F., Beer, J. S., & Klein, S. B. (2013). Self and identity as memory. The Handbook of Self and Identity, 68-90.
- [Background] Klein SB. Self, memory, and the self-reference effect: an examination of conceptual and methodological issues. Pers Soc Psychol Rev. 2012 Aug;16(3):283-300. doi: 10.1177/1088868311434214. Epub 2012 Jan 30. PMID 22291045
- [Background] Lancaster, S. L., & P. Hart, R. (2015). Military identity and psychological functioning: A pilot study. Military Behavioral Health, 3(1), 83-87. http://doi.org/10.1080/21635781.2014.995254
- [Background] Markus, H. (1977). Self-schemata and processing information about the self. Journal of Personality and Social Psychology, 35(2), 63-78.
- [Background] Markus, H., Crane, M., Bernstein, S., & Siladi, M. (1982). Self-schemas and gender. Journal of Personality and Social Psychology. http://doi.org/10.1037/0022-3514.42.1.38
- [Background] Markus, H., Hamill, R., & Sentis, K. P. (1987). Thinking fat: Self-schemas for body weight and the processing of weight relevant information. Journal of Applied Social Psychology, 17(1), 50-71. http://doi.org/10.1111/j.1559-1816.1987.tb00292.x
- [Background] Mayring, P. (2014). Qualitative content analysis. Theoretical foundation, basic procedures and software solution. Advances in Bioethics. http://doi.org/10.1016/S1479-3709(07)11003-7
- [Background] McNally RJ, Lasko NB, Macklin ML, Pitman RK. Autobiographical memory disturbance in combat-related posttraumatic stress disorder. Behav Res Ther. 1995 Jul;33(6):619-30. doi: 10.1016/0005-7967(95)00007-k. PMID 7654154
- [Background] Migliore, L. A., & Nathan, D. (2018) The Military Identity Project: Self-descriptive content and response time as indicators for presence of military self-schemas. Manuscript submitted for publication.
- [Background] Migliore, L. A., & Pound, L. B. (2016). The Military Identity Project: A mixed method investigation of military self-schema content. Military Behavioral Health, 4(2), 183-192. http://doi.org/10.1080/21635781.2015.1133351
- [Background] Noureddine S, Stein K. Healthy-eater self-schema and dietary intake. West J Nurs Res. 2009 Mar;31(2):201-18. doi: 10.1177/0193945908327157. Epub 2008 Dec 2. PMID 19050230
- [Background] Oyserman, D., Smith, G. C., & Elmore, K. C. (2014). Identity-based motivation: Implications for health and health disparities. Journal of Social Issues, 70(2), 206-225. http://doi.org/10.1111/josi.12056
- [Background] Rivers FM, Gordon S, Speraw S, Reese S. U.S. Army nurses' reintegration and homecoming experiences after Iraq and Afghanistan. Mil Med. 2013 Feb;178(2):166-73. doi: 10.7205/milmed-d-12-00279. PMID 23495462
- [Background] Ryff, C. D. (1989). Happiness is everything, or is it? Explorations on the meaning of psychological well-being. Journal of Personality and Social Psychology, 57(6), 1069.
- [Background] Ryff CD, Keyes CL. The structure of psychological well-being revisited. J Pers Soc Psychol. 1995 Oct;69(4):719-27. doi: 10.1037//0022-3514.69.4.719. PMID 7473027
- [Background] Scannell-Desch E, Doherty ME. Experiences of U.S. military nurses in the Iraq and Afghanistan wars, 2003-2009. J Nurs Scholarsh. 2010 Mar;42(1):3-12. doi: 10.1111/j.1547-5069.2009.01329.x. PMID 20487181
- [Background] Schaefer SM, Morozink Boylan J, van Reekum CM, Lapate RC, Norris CJ, Ryff CD, Davidson RJ. Purpose in life predicts better emotional recovery from negative stimuli. PLoS One. 2013 Nov 13;8(11):e80329. doi: 10.1371/journal.pone.0080329. eCollection 2013. PMID 24236176
- [Background] Smith, R., & True, G. (2014). Warring Identities: Identity conflict and the mental distress of American Veterans of the wars in Iraq and Afghanistan. Society and Mental Health. http://doi.org/10.1177/2156869313512212
- [Background] Stein, K. (1994). Complexity of the self-schema and responses to disconfirming feedback. Cognitive Therapy and Research, 18(2), 161-178. http://doi.org/10.1007/BF02357222
- [Background] Stein KF. The organizational properties of the self-concept and instability of affect. Res Nurs Health. 1995 Oct;18(5):405-15. doi: 10.1002/nur.4770180506. PMID 7676074
- [Background] Stein KF. The self-schema model: a theoretical approach to the self-concept in eating disorders. Arch Psychiatr Nurs. 1996 Apr;10(2):96-109. doi: 10.1016/s0883-9417(96)80072-0. PMID 8935986
- [Background] Stein KF, Corte C. Reconceptualizing causative factors and intervention strategies in the eating disorders: a shift from body image to self-concept impairments. Arch Psychiatr Nurs. 2003 Apr;17(2):57-66. doi: 10.1053/apnu.2003.50000. PMID 12701083
- [Background] Stein KF, Corte C. The identity impairment model: a longitudinal study of self-schemas as predictors of disordered eating behaviors. Nurs Res. 2008 May-Jun;57(3):182-90. doi: 10.1097/01.NNR.0000319494.21628.08. PMID 18496104
- [Background] Stein KF, Corte C, Chen DG, Nuliyalu U, Wing J. A randomized clinical trial of an identity intervention programme for women with eating disorders. Eur Eat Disord Rev. 2013 Mar;21(2):130-42. doi: 10.1002/erv.2195. Epub 2012 Sep 27. PMID 23015537
- [Background] Stein KF, Keller C, Corte C. Creando Posibilidades: A Cognitive Model of Risk Behaviors in Mexican American Women. J Food Nutr Disord. 2014 Jun;3(3):144. doi: 10.4172/2324-9323.1000144. Epub 2014 Jun 13. PMID 29911123
- [Background] Stein, K. F., & Nyquist, L. (2001). Disturbances in the self : A source of eating disorders. Eating Disorders Review, 12(1), 1-8.
- [Background] Stein KF, Roeser R, Markus HR. Self-schemas and possible selves as predictors and outcomes of risky behaviors in adolescents. Nurs Res. 1998 Mar-Apr;47(2):96-106. doi: 10.1097/00006199-199803000-00008. PMID 9536193
- [Background] Swann, W. B., & Bosson, J. K. (2010). Self and Identity. In Handbook of Social Psychology (pp. 589-628).
- [Background] ZAJONC RB. The process of cognitive tuning in communication. J Abnorm Soc Psychol. 1960 Sep;61:159-67. doi: 10.1037/h0047987. No abstract available. PMID 13787720